CLINICAL TRIAL: NCT04560296
Title: Community-based E-Health Program for Older Adults Living with Chronic Diseases - a Cluster Controlled Study with Process Evaluation
Brief Title: Community-based E-Health Program for Older Adults Living with Chronic Diseases
Acronym: CeHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Assistant Professor, National University of Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUHSRO/2019/081/Startup/06
Record Dates: First submitted 2020-09-03; First posted 2020-09-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemias
Keywords: community-dwelling older adults; chronic diseases; self-management; e-health; cognitive impairment
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Chronic Disease; Cognitive Dysfunction | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: Cluster Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community-based E-Health Program (Experimental): The intervention group will consist of 80 participants who will engage in Community-based E-Health Program.
  Interventions: Behavioral: Community-based E-Health Program
- usual self-management and follow up with doctors/nurse (Active Comparator): The participants will receive the usual self-management and follow up with doctors/nurse as planned.
  Interventions: Behavioral: usual self-management and follow up with doctors/nurse

INTERVENTIONS:
Behavioral: Community-based E-Health Program — Community-based E-Health Program will be developed to engage and empower older adults to manage the chronic conditions effectively.
  Arms: Community-based E-Health Program
Behavioral: usual self-management and follow up with doctors/nurse — usual self-management and follow up with doctors/nurse as planned in the community nurse post.
  Arms: usual self-management and follow up with doctors/nurse

SUMMARY:
With increased aging population, there is a higher rate of having chronic diseases and cognitive impairment. In order to achieve successful aging, it is important for community-dwelling older adults to perform better self-management with improved health literacy and various kinds of support. The study aims to develop a Community-based E-Health Program (CeHP) for Older Adults Living with Chronic Diseases , evaluate the effectiveness of CeHP, and refine the program based on the outcome measurement. A cluster controlled trial will be adopted. A follow-up process evaluation will be conducted to assess the acceptability, strengths and limitations of CeHP based on the participants' perspectives. The research contributes to engage and empower older adults living in the community to manage their chronic condition, and foster collaboration with the goal of translating evidence into action.

DETAILED DESCRIPTION:
Background:

With increased aging population, there is a higher rate of having chronic diseases and cognitive impairment. In order to achieve successful aging, it is important for community-dwelling older adults to perform better self-management with improved health literacy and various kinds of support.

Objectives:

The study aims to develop a Community-based E-Health Program (CeHP), evaluate the effectiveness of CeHP, and refine the program based on the outcome measurement.

Method:

The research team will develop the Community-based E-Health Program, and assess the effects of the program. A needs assessment will be carried out using focus group discussion with the older adults. A cluster controlled trial will be adopted. A follow-up process evaluation will be conducted to assess the acceptability, strengths and limitations of Community-based E-Health Program based on the participants' perspectives

Discussion and conclusion:

The proposed research contributes to engage and empower older adults living in the community to manage their chronic condition, and foster collaboration with the goal of translating evidence into action. This research will offer important insights into the need for educating and engaging older adults in managing chronic conditions to promote health and well-being, and therefore contribute to health and well-being of the elderly population.

ELIGIBILITY:
Inclusion Criteria:

1) aged 60 or above; 2) able to understand and communicate in either English or Mandarin; 3) able to give consent to participate; 4) lives within the community setting; 5) diagnosed with chronic conditions (Hypertension, Hyperlipidemia, and Diabetes Mellites); 6) able to commit to the research program throughout the whole duration.

Exclusion Criteria:

1. severe cognitive impairment;
2. severe psychiatric disorders;
3. severe vision impairment;
4. severe hearing impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Self-care ability of Chronic disease | baseline, 3 month, 6 month
  Self-care of Chronic Illness Inventory

SECONDARY OUTCOMES:
Change in Patient Empowerment | baseline, 3 month, 6 month
  Patient Empowerment scale
Change in Health Literacy | baseline, 3 month, 6 month
  Health Literacy Scale, minimum value is 12, maximum value is 48, higher scores mean a better outcome.
Change in Social support | baseline, 3 month, 6 month
  Social support Questionnaire
Change in Healthy Aging practice | baseline, 3 month, 6 month
  Healthy Aging Instrument
Montreal Cognitive Assessment | baseline, 3 month, 6 month
  Singapore version 2010
Symbol Digit modality test | baseline, 3 month, 6 month
  Quickly screens for organic cerebral dysfunction in both children and adults, patient substitutes a number, either orally or written, for randomized presentations of geometric figures
HbA1c | baseline, 3 month
  glycemic control
Lipid panel | baseline, 3 month
  HDL, LDL, triglycerides
Immunological profile | baseline, 3 month
  Cytokines (IL-1, IL6, IL15), TNFa, C1q, antinuclear antibody, antiDNA antibody
Hormones | baseline, 3 month
  Cortisol, DHEA, insulin
Fasting glucose | baseline, 3 month
  Plasma glucose concentration after fasting for 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Xi Wu, PhD, Principal Investigator — National University of Singapore
Locations (9):
- Singapore (9):
  - Brahm Centre @ Tampines, Singapore, Singapore
  - THK SAC @ Bedok Radiance, Singapore
  - THK SAC @ Kaki Bukit, Singapore
  - Pap Community Foundation 3-in-1 Family Centre (Aged Care), Singapore
  - Brahm Centre @ Simei 227, Singapore
  - Lb Sac @ 434 Tampines, Singapore
  - Presbyterian Community Services - Evergreen Circle Seniors Activity Centre, Singapore
  - Lb Sac @ 499C Tampines, Singapore
  - Lb Sac (Sa) @ Tampines 494E, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epidemiology & Disease Control Division, et al., The Burden of Disease in Singapore, 1990-2017: An overview of the Global Burden of Disease Study 2017results. 2019: Seattle, WA: IHME
- [Background] van der Heide I, Poureslami I, Mitic W, Shum J, Rootman I, FitzGerald JM. Health literacy in chronic disease management: a matter of interaction. J Clin Epidemiol. 2018 Oct;102:134-138. doi: 10.1016/j.jclinepi.2018.05.010. Epub 2018 May 21. PMID 29793001
- [Background] Vijayan M, Reddy PH. Stroke, Vascular Dementia, and Alzheimer's Disease: Molecular Links. J Alzheimers Dis. 2016 Sep 6;54(2):427-43. doi: 10.3233/JAD-160527. PMID 27567871
- [Background] Tan HH, Xu J, Teoh HL, Chan BP, Seet RC, Venketasubramanian N, Sharma VK, Chen CL, Dong Y. Decline in changing Montreal Cognitive Assessment (MoCA) scores is associated with post-stroke cognitive decline determined by a formal neuropsychological evaluation. PLoS One. 2017 Mar 27;12(3):e0173291. doi: 10.1371/journal.pone.0173291. eCollection 2017. PMID 28346532
- [Background] van de Bovenkamp HM, Dwarswaard J. The complexity of shaping self-management in daily practice. Health Expect. 2017 Oct;20(5):952-960. doi: 10.1111/hex.12536. Epub 2017 Feb 2. PMID 28152248
- [Background] Koetsenruijter J, van Eikelenboom N, van Lieshout J, Vassilev I, Lionis C, Todorova E, Portillo MC, Foss C, Serrano Gil M, Roukova P, Angelaki A, Mujika A, Knutsen IR, Rogers A, Wensing M. Social support and self-management capabilities in diabetes patients: An international observational study. Patient Educ Couns. 2016 Apr;99(4):638-643. doi: 10.1016/j.pec.2015.10.029. Epub 2015 Nov 2. PMID 26549171
- [Background] Beauchamp A, Peeters A, Tonkin A, Turrell G. Best practice for prevention and treatment of cardiovascular disease through an equity lens: a review. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):599-606. doi: 10.1097/HJR.0b013e328339cc99. PMID 20562629
- [Background] Solomon M, Wagner SL, Goes J. Effects of a Web-based intervention for adults with chronic conditions on patient activation: online randomized controlled trial. J Med Internet Res. 2012 Feb 21;14(1):e32. doi: 10.2196/jmir.1924. PMID 22353433